CLINICAL TRIAL: NCT00420186
Title: A Phase I Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of BMS-690514 in Combination With Paclitaxel and Carboplatin for Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study of BMS-690514 in Combination With Paclitaxel and Carboplatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA187-004
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2014-05

CONDITIONS: Cancer (Solid Tumors)
MeSH Terms: conditions — Neoplasms | interventions — BMS-690514

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: BMS-690514

INTERVENTIONS:
Drug: BMS-690514 — Tablets / IV, Oral / IV, 100 to 300 mg / Paclitaxel (200 mg/m2) / Carboplatin dose (mg) = Target AUC (6) x (GFR + 25), Once daily Days 4-19, up to 24 mos
  Other Names: panHER

SUMMARY:
The purpose of this clinical research is to assess the safety and tolerability of BMS-690514 when given in combination with paclitaxel and carboplatin. Paclitaxel and carboplatin will be administered on a standard regimen every 3 weeks at standard doses. BMS-690514 will be given in the interval at escalating doses until the maximum tolerated dose (MTD) is identified. An additional cohort of subjects will be treated with BMS-690514 at the MTD in combination with Paclitaxel and carboplatin

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic solid tumors for whom paclitaxel/carboplatin is considered an appropriate therapy
* Centrally located squamous cell carcinoma of the lung is permitted
* ECOG performance status of 0-1
* Life expectancy of at least 3 months
* Men and women age 18 and above

Exclusion Criteria:

* Symptomatic brain metastases. Patients with signs for symptoms of brain metastases are ineligible unless brain metastases are ruled out by CT or MRI
* Peripheral neuropathy ≥Grade 1 for any reason
* History of thromboembolic disease or bleeding diatheses within the last 6 months
* Women of child bearing potential without adequate contraception, breastfeeding, or pregnant
* Serious, uncontrolled medical disorder or active infection
* Uncontrolled or significant cardiac disease
* Uncontrolled hypertension (150/100)
* Allergy to Cremophor EL®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability and to identify a dose for BMS-690514 in combination with paclitaxel/carboplatin for Phase II evaluation | upon occurrence

SECONDARY OUTCOMES:
Describe anti-tumor activity | upon occurence
Obtain blood, plasma and fresh and/or archived tumor tissue for exploratory research | upon occurence

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
- Local Institution, Ottawa, Ontario, Canada
- Local Institution, Manchester, Greater Manchester, United Kingdom

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx